CLINICAL TRIAL: NCT02151240
Title: A Multi-centered, Randomized Study to Evaluate the Efficacy and Safety of Foscarnet Sodium and Sodium Chloride Injection Compared to Intravenous Acyclovir in Patients With Herpes Zoster From China
Brief Title: Efficacy and Safety of Foscarnet Sodium and Sodium Chloride Injection in Patients With Herpes Zoster
Acronym: Focus-101
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cttq (Industry)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cttq-focus-101
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2021-06-28 (Actual); Status verified 2021-06

CONDITIONS: Herpes Zoster
Keywords: herpes zoster, Foscarnet Sodium, Acyclovir, Postherpetic neuralgia
MeSH Terms: conditions — Herpes Zoster; Neuralgia, Postherpetic | interventions — Foscarnet; Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Foscarnet Sodium and Sodium Chloride Injection 3g: 250ml, IV; Second administration: Foscarnet Sodium and Sodium Chloride Injection 3g: 250ml, IV
  Interventions: Drug: Foscarnet Sodium
- Arm II (Active Comparator): First administration: Acyclovir for Injection 0.25g + 0.9% Sodium Chloride Injection 250ml, IV; Acyclovir for Injection 0.25g + 0.9% Sodium Chloride Injection 250ml, IV; Second administration: Acyclovir for Injection 0.25g+ 0.9% Sodium Chloride Injection 250ml, IV
  Interventions: Drug: Acyclovir

INTERVENTIONS:
Drug: Foscarnet Sodium
  Arms: Arm I
Drug: Acyclovir
  Arms: Arm II

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Foscarnet Sodium and Sodium Chloride Injection in patients with herpes zoster, and observe incidence of Postherpetic neuralgia

ELIGIBILITY:
Inclusion Criteria:

1.Patients with clinical diagnosis of Herpes Zoster, and able to be enrolled into the study ≤ 72 hours from appearance of rash; 2.18-65 years old, men and women; 3.VAS score≥4; 4.Patients haven't receive any antiviral medication before enrollment; 5.Patients able to understand the study procedures, agree to participate and give written consent.

Exclusion Criteria:

1. Patients with history of allergy to Foscarnet Sodium or Acyclovir;
2. Other combined infection (bacteria, fungi)
3. Severe decline in immune function, or long-term use of corticosteroid and immunosuppressor
4. Serious liver or renal function abnormalities (Aspartate Transaminase(AST) or alanine transaminase(ALT) ≥ 2.5x upper limits of normal(ULN), Creatinine(Cr) or Blood urea nitrogen(BUN)≥ 1x ULN)
5. Women who are pregnant or lactating, and women of childbearing potential failed to use an adequate method of contraception to avoid pregnancy;
6. Patients using other antiviral drugs;
7. Long-term use of non-steroid anti-inflammatory drug, tricyclic antidepressant, anti-epileptic drugs or analgesic
8. Current malignant tumor;
9. Patients investigators consider as inappropriate to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-05; Primary Completion 2015-05 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Effective rate | 8th days
  Effective rate = (No. of patients achieving recovery+ markedly improvement)/Total patients No.×100%.
  Recovery: curative index≥90%; Markedly improved: curative index 60%-89%; Improved: curative index 20%-59%; Ineffective: curative index<20%. Where Curative Index= (patient's pre-treatment condition score - post-treatment condition score)/pre-treatment condition score ×100%

SECONDARY OUTCOMES:
Incidence of Postherpetic neuralgia | 3rd month
number of participants with adverse event and serious adverse event | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Result] Breton G, Fillet AM, Katlama C, Bricaire F, Caumes E. Acyclovir-resistant herpes zoster in human immunodeficiency virus-infected patients: results of foscarnet therapy. Clin Infect Dis. 1998 Dec;27(6):1525-7. doi: 10.1086/515045. PMID 9868672
- [Result] Safrin S, Berger TG, Gilson I, Wolfe PR, Wofsy CB, Mills J, Biron KK. Foscarnet therapy in five patients with AIDS and acyclovir-resistant varicella-zoster virus infection. Ann Intern Med. 1991 Jul 1;115(1):19-21. doi: 10.7326/0003-4819-115-1-19. PMID 1646585